CLINICAL TRIAL: NCT06104124
Title: A Phase 3 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Dazodalibep in Participants With Sjögren's Syndrome With Moderate-to-severe Systemic Disease Activity
Brief Title: A Study to Evaluate the Efficacy and Safety of Dazodalibep in Participants With Sjögren's Syndrome (SS) With Moderate-to-severe Systemic Disease Activity
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HZNP-DAZ-301; 2023-503904-10-00 (Registry Identifier: EU Clinical Trial Information System)
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Sjogren's Syndrome
Keywords: Sjögren's Syndrome With Moderate-to-severe Systemic Disease Activity Study Phase: Phase 3; European Alliance of Associations for Rheumatology Sjögren's Syndrome Disease Activity Index (ESSDAI); European Alliance of Associations for Rheumatology Sjögren's Syndrome Patient Reported Index (ESSPRI); European Alliance of Associations for Rheumatology (EULAR)
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dazodalibep Dose 1 (Experimental): Participants will be administered dose 1 of dazodalibep by intravenous (IV) infusion.
  Interventions: Drug: Dazodalibep
- Dazodalibep Dose 2 (Experimental): Participants will be administered dose 2 of dazodalibep by IV infusion.
  Interventions: Drug: Dazodalibep
- Placebo (Placebo Comparator): Participants will be administered placebo by IV infusion.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dazodalibep — IV infusion
  Other Names: VIB 4920; MEDI 4920
  Arms: Dazodalibep Dose 1; Dazodalibep Dose 2
Drug: Placebo — IV infusion
  Arms: Placebo

SUMMARY:
Primary Objective:

To evaluate the effect of dazodalibep on systemic manifestations of Sjögren's Syndrome (SS) in participants with moderate-to-severe systemic disease activity.

Secondary Objectives:

1. To evaluate the effect of dazodalibep on patient reported outcomes (PROs) in participants with SS.
2. To evaluate the safety and tolerability of dazodalibep in participants with SS

DETAILED DESCRIPTION:
Acquired from Horizon in 2024.

ELIGIBILITY:
Key Inclusion Criteria:

* Diagnosed with Sjögren's syndrome (SS) by meeting the 2016 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology (EULAR) Classification Criteria.
* Have an European Alliance of Associations for Rheumatology Sjögren's Syndrome Disease Activity Index (ESSDAI) score of >= 5 despite symptomatic or local therapy at screening.
* Positive for either anti-Ro autoantibodies or rheumatoid factor (RF), or both at screening (as per the central laboratory test).

Key Exclusion Criteria:

* Medical history of confirmed deep vein thrombosis, pulmonary embolism, or arterial thromboembolism within 2 years of screening.
* Active malignancy or history of malignancy within the last 5 years, except in situ carcinoma of cervix treated with apparent success with curative therapy > 12 months prior to screening OR cutaneous basal cell carcinoma following presumed curative therapy.
* Individuals with any severe or life-threatening cardiovascular (including vasculitis), respiratory, endocrine, gastrointestinal, hematological, psychiatric, or systemic disorder or any other condition that would place the individual at unacceptable risk of complications, interfere with evaluation of the IP, or confound the interpretation of participant safety or study results.
* Individuals who have a positive test for hepatitis B, hepatitis C, or HIV infection. A positive test for hepatitis B at screening is defined as: (1) positive for HBsAg OR (2) positive for either HBcAb or HBsAb and HBV DNA detected above the LLOQ by reflex testing by the central laboratory at screening.
* Active TB or untreated (per local guidelines) latent TB
* Individuals with a history of more than one episode of herpes zoster and/or any opportunistic infection in the last 12 months, and active infection requiring systemic treatment at the time of screening or through randomization, or history of more than 2 infections requiring intravenous (IV) antibiotics within 12 months prior to screening.
* Individuals who have received a live (attenuated) vaccine within the 4 weeks prior to randomization or plan to receive a live vaccine during their participation in the study.
* Last administration of experimental or investigational biologic or oral agents < 6 months prior to screening.
* Individuals who have had previous treatment with any biologic B-cell-depleting therapy (eg, rituximab, ocrelizumab, inebilizumab, ofatumumab, or ianalumab) within 12 months or other B-cell-targeting therapy (eg, belimumab) < 3 months prior to screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 651 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2026-08-19 (Estimated); Study Completion 2026-08-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in European Alliance of Associations for Rheumatology Sjögren's Syndrome Disease Activity Index (ESSDAI) Score | At Week 48

SECONDARY OUTCOMES:
Proportion of participants achieving ESSDAI response | At Week 48
Change from baseline in Diary for Assessing Sjogren's Patient-Reported Outcome Index (DASPRI) dryness domain score | At Week 48
Change from baseline in ESSPRI dryness domain score | At Week 48
Change from baseline in DASPRI dryness domain score | At Week 48
Change from baseline in tender and swollen joint counts | At Week 48
Change from baseline in Patient-Reported Outcomes Measurement Information System Fatigue-Short Form 10a (PROMIS-Fatigue-SF-10a) | At Week 48
Change from baseline in ESSDAI score | Week 12 and Week 24
Change from baseline in DASPRI total score | At Week 48
Change from baseline in ESSPRI total score | At Week 48
Change from baseline in total stimulated salivary flow | At Week 48
Number of participants With Treatment Emergent Adverse Events (TEAEs) | Baseline (Day 1) to Week 56
Number of participants With Treatment Emergent Serious Adverse Events (TESAEs) | Up to Week 56
Number of participants With Adverse Events of Special Interest (AESIs) | Up to Week 56

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (216):
- United States (45):
  - Arizona Arthritis & Rheumatology Associates - Avondale, Avondale, Arizona
  - Arizona Research Clinic PLLC, Chandler, Arizona
  - Arizona Arthritis and Rheumatology Associates - Flagstaff - 399 S Malpais Ln, Flagstaff, Arizona
  - Arizona Arthritis and Rheumatology Associates - Gilbert - 3645 S Rome St, Gilbert, Arizona
  - Arizona Arthritis and Rheumatology Associates - Glendale - 5681 W Beverly Ln, Glendale, Arizona
  - Arizona Arthritis and Rheumatology Associates - Tucson - 2001 W Orange Grove Rd, Tucson, Arizona
  - UCSD Altman Clinical and Translational Research Institute Building, La Jolla, California
  - Inland Rheumatology Clinical Trials Incorporated, Upland, California
  - Tekton Research, LLC - 2121 E Harmony Rd - PPDS, Fort Collins, Colorado
  - Bradenton Research Center Inc, Bradenton, Florida
  - Clinical Research of West Florida Inc - Clearwater, Clearwater, Florida
  - University of Miami - Leonard M. Miller School of Medicine, Miami, Florida
  - Suncoast Clinical Research - ATLAS - New Port Richey - PPDS, New Port Richey, Florida
  - Millennium Research, Ormond Beach, Florida
  - West Broward Rheumatology Associates, Inc., Tamarac, Florida
  - BayCare Medical Group, Tampa, Florida
  - Augusta University Medical Center-Augusta-1120 15th St, Augusta, Georgia
  - OrthoIllinois, LTD, Rockford, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Massachusetts General Hospital, Boston, Massachusetts
  - Clinical Research Institute of Michigan, LLC-St. Claire Shores, Saint Clair Shores, Michigan
  - Kansas City Physician Partners-8350 N Saint Clair Ave, Kansas City, Missouri
  - Arthritis, Rheumatic & Bone Disease Associates - P, Voorhees Township, New Jersey
  - NYU Langone Health - Joseph S. and Diane H. Steinberg Ambulatory Care Center, Brooklyn, New York
  - Arthritis and Osteoporosis Consultants of The Carolinas - Charlotte - 1918 Randolph Rd, Charlotte, North Carolina
  - Duke Early Phase Clinical Research Unit - PPDS, Durham, North Carolina
  - Onsite Clinical Solutions, LLC - Salisbury, Salisbury, North Carolina
  - Arthritis & Osteoporosis Center of Southwest Ohio - Miamisburg, Miamisburg, Ohio
  - University of Toledo Medical Center, Toledo, Ohio
  - STAT Research-600 Aviator Ct, Vandalia, Ohio
  - Low Country Rheumatology PA-Summerville, Summerville, South Carolina
  - Murfreesboro Medical Clinic Westlawn, Murfreesboro, Tennessee
  - Amarillo Center For Clinical Research, Amarillo, Texas
  - Tekton Research, LLC - W Gate Blvd - Austin - PPDS, Austin, Texas
  - Accurate Clinical Management-Baytown, Baytown, Texas
  - Precision Comprehensive Clinical Research Solutions, Grapevine, Texas
  - Prolato Clinical Research Center, Houston, Texas
  - R & H Clinical Research-777 S Fry Rd, Katy, Texas
  - Valley Arthritis Center, McAllen, Texas
  - University of Texas - San Antonio - Health Science Center - PPDS, San Antonio, Texas
  - DM Clinical Research - Migraine and COPD - PPDS, Tomball, Texas
  - Metrodora Institute, West Valley City, Utah
  - Overlake Arthritis & Osteoporosis Center, Bellevue, Washington
  - Western Washington Medical Group, Bothell - Rheumatology, Bothell, Washington
  - Rheumatology and Pulmonary Clinic, Beckley, West Virginia
- Argentina (17):
  - Sanatorio Agote - Swiss Medical Group - PPDS, Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Framingham Centro Médico, La Plata, Buenos Aires
  - Instituto CER S.A., Quilmes, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes SRL, Quilmes, Buenos Aires
  - MR Medicina Reumatologica, San Fernando, Buenos Aires
  - Hospital General de Agudos Dr. José María Ramos Mejia, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Expertia S.A- Mautalén Salud e Investigación, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Centro Privado de Medicina Familiar, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Consultorios Médicos Dr. Doreski - Fundacion Respirar - PPDS, Buenos Aires, Ciudad Autónoma de BuenosAires
  - Sanatorio Allende S.A, Córdoba, Córdoba Province
  - Centro de Investigaciones Médicas Tucumán - PPDS, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Reumatológicas, San Miguel de Tucumán, Tucumán Province
  - Clínica Mayo de U.M.C.B. S.R.L, San Miguel de Tucumán, Tucumán Province
  - DOM Centro de Reumatología, Buenos Aires
  - Aprillus Asistencia e Investigacion de Arcis Salud SRL, Buenos Aires
  - Centro Medico Arsema, Buenos Aires
  - Centro Polivalente de Asistencia e Investigación Clínica - CER San Juan, San Juan
- The Queen Elizabeth Hospital, Woodville South, South Australia, Australia
- Belgium (2):
  - UZ Gent, Ghent, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
- Brazil (6):
  - SER - Serviços Especializados em Reumatologia da Bahia S/S - ME, Salvador, Estado de Bahia
  - AES - AS - L2IP - Instituto de Pesquisas Clínicas LTDA Brasilia, Brasília, Federal District
  - Irmandade da Santa Casa de Misericórdia de Belo Horizonte - PPDS, Belo Horizonte, Minas Gerais
  - Centro Mineiro de Pesquisa - CMiP, Juiz de Fora, Minas Gerais
  - Centro de Estudos em Terapias Inovadoras, Curitiba, Paraná
  - LMK Servicos Medicos SS, Porto Alegre, Rio Grande do Sul
- Centre de Recherche Musculo-Squelettique - 1920 Rue Bellefeuille, Trois-Rivières, Quebec, Canada
- Chile (5):
  - Clinical Research Chile SpA - PPDS, Valdivia, Los Ríos Region
  - Centro de especialidades médicas Vanguardia, Temuco, Región de la Araucanía
  - Centro de Investigacion de Enfermedades Respiratorias e inmunologicas, Viña del Mar, Región de Valparaíso
  - Enroll SpA - Dr. Manuel Barros Borgono - PPDS, Providencia, Región-MetropolitanadeSantiago
  - BIOCINETIC Ltda, Santiago, Región-MetropolitanadeSantiago
- Croatia (4):
  - Clinical Center Zagreb - Oncology - Salata 7 - PPDS, Zagreb, City of Zagreb
  - Polyclinic Bonifarm, Zagreb, City of Zagreb
  - Clinical Hospital Centre Osijek, Osijek
  - University Hospital of Split-Spinciceva 1, Split
- France (5):
  - Hopital Emile Muller, Mulhouse, Haut-Rhin
  - CHU de Bordeaux - Hôpital Saint-André, Bordeaux
  - CHU de Brest - Hôpital La Cavale Blanche, Brest
  - AP-HP - Hôpital Bicêtre, Le Kremlin-Bicêtre
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
- Germany (4):
  - Rheumazentrum Prof. Dr. med. Gunther Neeck-Standort Bad Doberan, Bad Doberan, Mecklenburg-Vorpommern
  - Rheumazentrum Greifswald, Greifswald Hansestadt, Mecklenburg-Vorpommern
  - DRK Gemeinnützige Krankenhaus GmbH Sachsen - DRK Krankenhaus Chemnitz-Rabenstein, Chemnitz
  - MVZ Rheuma, Hamburg
- Greece (5):
  - Olympion General Clinic, Kato Sychena Patras, Achaïa
  - Naval Hospital of Athens, Athens, Attica
  - Laiko General Hospital of Athens, Athens, Attica
  - University General Hospital of Larissa, Larissa, Larisa
  - Euromedica Kianous Stavros, Thessaloniki
- Hungary (4):
  - Bekes Varmegyei Kozponti Korhaz, Gyula, Bekes County
  - Vasarhelyi Sarkanyfu Kft., Hódmezővásárhely, Csongrád megye
  - Debreceni Egyetem Klinikai Kozpont Nagyerdei Campus, Debrecen, Hajdú-Bihar
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet - Albert Flórián út 5-7, Budapest
- Israel (2):
  - Meir Medical Center, Kfar Saba, Central District
  - The Chaim Sheba Medical Center - PPDS, Ramat Gan
- Italy (10):
  - AUSL di Reggio Emilia - IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia, Emilia-Romagna
  - Azienda Sanitaria Universitaria Friuli Centrale - PO Universitario Santa Maria della Misericordia, Udine, Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Fondazione Policlinico Universitario A Gemelli - Rome - PPDS, Rome, Lazio
  - Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Lombardy
  - A.O.U. Città della Salute e della Scienza di Torino, Turin, Piedmont
  - AOU Policlinico Gaspare Rodolico-San Marco - Presidio Ospedaliero San Marco, Catania, Sicily
  - Azienda Ospedaliera Universitaria Careggi, Florence, Tuscany
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento Santa Chiara, Pisa, Tuscany
  - Azienda Ospedaliera Universitaria Integrata Di Verona, Verona, Veneto
- Japan (23):
  - Chubu Rosai Hospital, Nagoya, Aiti
  - Japan Community Health Care Organization (JCHO) Chukyo Hospital, Nagoya, Aiti
  - Daido Clinic, Nagoya, Aiti
  - Sapporo Medical University Hospital, Sapporo, Hokkaidô
  - Hokkaido University Hospital, Sapporo, Hokkaidô
  - Hospital of the University of Occupational and Environmental Health, Japan, Kita Kyushu-shi, Hukuoka
  - Hyogo Medical University Hospital, Nishinomiya-Shi, Hyôgo
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Kanazawa Medical University Hospital, Kahoku, Ishikawa-ken
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - National Hospital Organization Yokohama Medical Center, Yokohama, Kanagawa
  - University Hospital, Kyoto Prefectural University of Medicine, Kyoto, Kyôto
  - Kyoto University Hospital, Kyoto, Kyôto
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Sasebo Chuo Hospital, Sasebo-Shi, Nagasaki
  - Kurashiki Medical Clinic, Kurashiki-Shi, Okayama-ken
  - Saitama Medical University Hospital, Iruma-gun, Saitama
  - Hamamatsu University Hospital, Hamamatsu, Shizuoka
  - Nippon Medical School Hospital, Bunkyo-Ku, Tokyo
  - St. Luke's International Hospital, Chuo-Ku, Tokyo
  - Tokyo Medical Center, Meguro-Ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Nihon University Itabashi Hospital, tabashi City, Tokyo
- Mexico (15):
  - Mediadvance Clinical S.A.P.I. de C.V., Parques de San Felipe, Chihuahua
  - ONCOR - Centro de Infusion e Investigación Oncologia de Saltillo S.C, Saltillo, Coahuila
  - CIMAB SA de CV, Torreón Centro, Coahuila
  - Centro de Investigación en Artritis y Osteoporosis - PPDS, Mexicali, Estado de Baja California
  - Centro de Estudios de Investigacion Basica Y Clinica SC, Guadalajara, Jalisco
  - Bioclinica - Centro Integral En Reumatologia Sociedad Anónima de Capital Variable - PPDS, Guadalajara, Jalisco
  - Cryptex Investigación Clínica, S.A. de C.V., Mexico City, Mexico City
  - Centro de Investigación y Tratamiento Reumatológico S.C, San Miguel Chapultepec, Mexico City
  - Unidad de Atencion Medica e Investigacion en Salud, Mérida, Yucatán
  - Centro de Investigacion Farmacologica Del Bajio Sc, León
  - Consultorio de Reumatologia, México
  - Clinstile, S.A. de C.V., México
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Mitras Centro
  - Accelerium, S. de R.L. de C.V. - PPDS, Monterrey
  - Oaxaca Site Management Organization - Clinic - OSMO - PPDS, Oaxaca City
- New Zealand (3):
  - Optimal Clinical Trials Ltd - PPDS, Auckland
  - Aotearoa Clinical Trials Trust, Auckland
  - Health New Zealand - Te Whatu Ora - Waikato (Waikato Hospital), Hamilton
- Peru (7):
  - Clinica San Antonio S.A.C, Trujillo, La Libertad
  - Clinica San Juan Bautista, San Juan de Lurigancho, Lima region
  - Hogar Clinica San Juan de Dios - Arequipa, Arequipa
  - Hospital Militar Central Luis Arias Schereiber, Lima
  - Clínica Internacional San Borja-Avenida Guardia Civil 385, Lima
  - Instituto de Ginecologia y Reproduccion - PPDS, Lima
  - Alfredo Berrocal Kasay Reuma Sociedad de Responsabilidad Limitada, Pueblo Libre
- Poland (28):
  - Pratia Poznan - PPDS, Poznan, Greater Poland Voivodeship
  - Med-Polonia Sp. z o.o., Poznan, Greater Poland Voivodeship
  - Prywatna Praktyka Lekarska Pawel Hrycaj, Poznan, Greater Poland Voivodeship
  - Malopolskie Centrum Kliniczne, Krakow, Lesser Poland Voivodeship
  - Centrum Medyczne Oporow, Wroclaw, Lower Silesian Voivodeship
  - Dolnoslaski Szpital Specjalistyczny im. T. Marciniaka, Centrum Medycyny Ratunkowej, Wroclaw, Lower Silesian Voivodeship
  - ETG Lublin - PPDS, Lublin, Lublin Voivodeship
  - Reumed Sp. z o.o., Lublin, Lublin Voivodeship
  - FutureMeds - Warszawa Centrum - PPDS, Warsaw, Masovian Voivodeship
  - MICS Centrum Medyczne Warszawa - MICS - PPDS, Warsaw, Masovian Voivodeship
  - MTZ Clinical Research Powered by PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Narodowy Instytut Geriatrii, Reumatologii i Rehabilitacji im. Prof. Dr hab. Med. Eleonory Reicher, Warsaw, Masovian Voivodeship
  - Klinika Reuma Park sp . zoo Sp.k., Warsaw, Masovian Voivodeship
  - FutureMeds - Targowek - PPDS, Warsaw, Masovian Voivodeship
  - K2J2 Medical Center, Wołomin, Masovian Voivodeship
  - Centrum Badawcze Panaceum Agnieszka Brzezicka Magdalena Lenkiewicz Sp. Z o.o., Malbork, Pomeranian Voivodeship
  - MICS Centrum Medyczne Bydgoszcz, Bydgoszcz
  - Szpital Uniwersytecki Nr 2 im. Dr Jana Biziela w Bydgoszczy, Bydgoszcz
  - Centrum Medyczne Pratia Katowice - PPDS, Katowice
  - Centrum Medyczne Plejady Magdalena Celinska - Lowenhoff, Michal Zolnowski Spolka komandytowa, Krakow
  - Centrum Medyczne PROMED- Olszanska 5G, Krakow
  - FutureMeds - Lodz - PPDS, Lodz
  - Twoja Przychodnia PCM, Poznan
  - ETG Warszawa - PPDS, Warsaw
  - WIM-PIB, Centralny Szpital Kliniczny MON, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza Radeckiego we Wroclawiu - Borowska 213, Wroclaw
  - Pracownia Badan Klinicznych Salus - ul. Ołtaszyńska 92c/3, Wroclaw
  - FutureMeds - Wroclaw - PPDS, Wroclaw
- Portugal (4):
  - ULS de Lisboa Ocidental, EPE - Hospital Egas Moniz, Lisbon, Lisbon District
  - Hospital Conde de Bertiandos - Unidade Local de saúde do Alto Minho, EPE - Ponte de Lima, Ponte de Lima, Viana do Castelo District
  - Centro Hospitalar Universitário Lisboa Norte, E.P.E - PPDS, Lisbon
  - ULS de Gaia/Espinho, EPE - Unidade I, Vila Nova de Gaia
- GCM Medical Group, PSC -62 Calle Jose Marti, San Juan, Puerto Rico
- Serbia (6):
  - Institute of Rheumatology - PPDS, Belgrade
  - Military Medical Academy, Belgrade
  - University Clinical Center of Serbia - Pasterova 2 - PPDS, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Centre of Vojvodina, Novi Sad
  - Special Hospital For Rheumatic Diseases Novi Sad, Novi Sad
- The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul, South Korea
- Spain (9):
  - C.H. Regional Reina Sofia - PPDS, Córdoba, Córdoba
  - Hospital Regional Universitario de Malaga - Hospital Civil, Málaga, Málaga
  - Hospital Universitario de Basurto, Bilbao
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Fundacio Hospital de l'Esperit Sant, Santa Coloma de Gramenet(Barcelona)
  - Hospital Universitario de Canarias, Santa Cruz de Tenerife
  - Hospital Quironsalud Infanta Luisa, Seville
  - Hospital Nuestra Señora de Valme, Seville
- Taiwan (4):
  - Chang Gung Memorial Hospital, Linkou, Gui Shan Qu
  - Kaohsiung Medical University - Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Taipei Medical University Hospital - PPDS, Taipei
- United Kingdom (4):
  - Chapel Allerton Hospital - PPDS, Leeds
  - William Harvey Research Institute - PPDS, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Queen Alexandra Hospital, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual patient data for variables necessary to address the specific research question in an approved data sharing request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data sharing requests relating to this study will be considered beginning 18 months after the study has ended and either 1) the product and indication have been granted marketing authorization in both the US and Europe or 2) clinical development for the product and/or indication discontinues and the data will not be submitted to regulatory authorities. There is no end date for eligibility to submit a data sharing request for this study.
Access Criteria: Qualified researchers may submit a request containing the research objectives, the Amgen product(s) and Amgen study/studies in scope, endpoints/outcomes of interest, statistical analysis plan, data requirements, publication plan, and qualifications of the researcher(s). In general, Amgen does not grant external requests for individual patient data for the purpose of re-evaluating safety and efficacy issues already addressed in the product labelling. Requests are reviewed by a committee of internal advisors. If not approved, a Data Sharing Independent Review Panel will arbitrate and make the final decision. Upon approval, information necessary to address the research question will be provided under the terms of a data sharing agreement. This may include anonymized individual patient data and/or available supporting documents, containing fragments of analysis code where provided in analysis specifications. Further details are available at the URL below.
URL: http://www.amgen.com/datasharing

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com